CLINICAL TRIAL: NCT05015556
Title: Minimal Invasive Volar Plating Versus Cast Immobilization for Treatment of Stable Non-displaced Distal Radial Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goorens Chul Ki (Other)
Responsible Party: Sponsor-Investigator, Goorens Chul Ki, M.D., Principal Investigator, Regionaal Ziekenhuis Heilig Hart Tienen
Organization: Regionaal Ziekenhuis Heilig Hart Tienen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109
Record Dates: First submitted 2021-06-03; First posted 2021-08-20 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Radius Fracture Distal
Keywords: Minimal invasive; Osteosynthesis; Conservative treatment; Cost effectiveness
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding of results by computer of the outcome results. Blinding of the patients or the care provider is not possible due to the obvious differences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Casting (No Intervention): Casting of the distal radius for 6 weeks
- Minimal invasive volar plating (Active Comparator): Muscle sparing osteosynthesis, no casting postoperatively
  Interventions: Procedure: Minimal invasive volar plating

INTERVENTIONS:
Procedure: Minimal invasive volar plating — Muscle sparing osteosynthesis, no casting postoperatively
  Arms: Minimal invasive volar plating

SUMMARY:
Nondisplaced distal radial fractures are nowadays treated by plaster cast immobilization. In this study, the investigators challenge this classical standard treatment with a surgical solution: minimal invasive volar plating with pronatus quadratus sparing approach. Potential benefits of this surgical treatment are higher cost effectiveness, economical benefit, earlier recuperation of professional and recreational activities, earlier functional recuperation by faster clinical recovery (range of motion, grip strength) and decreased risk of secondary fracture displacement. Potential drawbacks are surgical risks and complications.

DETAILED DESCRIPTION:
Randomized controlled trial Number still to be determined by power analysis on economical outcome measurement Similar study number = 90 Randomization by computer.

RZ Tienen, Dr Goorens Level 4 hand surgeon

Inclusion criteria:

* Stable distal radial fractures (volar tilt <10° dorsal tilt, <2mm impaction, <2mm articular depression)
* 18 - 65 years, professional active

Exclusion criteria:

* associated lesions, open fractures, unstable, displaced fractures
* neurological disorder affecting the upper limb, history of wrist lesion involving the same wrist, dementia, substance abuse, severe psychiatric disorder and previous injured contralateral wrist

Treatment

1. Cast treatment: 6 weeks with 1 plaster exchange of after 2 weeks
2. Minimal invasive plating: no cast

Followup 2 weeks, 6 weeks, 3 months, 6 months, 1 year

Primary PROM:

* Cost effectiveness: QALY SF-36
* Direct costs: surgery, hospitalisation, follow-up consultations, imaging, medication, wound care, nurse cost, physiotherapy cost
* Indirect costs: loss of productivity (SF-HLQ)
* Health insurances costs
* Confounding factors

  * Independent vs servant
  * Insurance?
  * Work type?
  * Age, sex, dominance
* Work absence, professional recuperation
* Recreational sport resumption

Secondary PROM

* ROM (F/E/RD/UD/P/S)
* Grip strength (Jamar)
* Pain (VAS)
* DASH scare, PRWE score
* Satisfaction (VAS), would you do it again?
* RX ulna variance, radial tilt
* complications

ELIGIBILITY:
Inclusion Criteria:

* Stable distal radial fractures (volar tilt <10° dorsal tilt, <2mm impaction, <2mm articular depression)
* 18 - 65 years, professional active

Exclusion Criteria:

* associated lesions, open fractures, unstable, displaced fractures
* neurological disorder affecting the upper limb, history of wrist lesion involving the same wrist, dementia, substance abuse, severe psychiatric disorder and previous injured contralateral wrist

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
QALY | 1 year
  Using the Short Form 36 (SF-36) assessment - cost effectiveness (The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.)
Costs | 1 year
  Direct, indirect, health insurances

SECONDARY OUTCOMES:
Wrist ROM | 1 year
  Range of motion (flexion, extension, radial deviation, ulnar deviation, pronation, supination)
Grip Strength | 1 year
  Using the Jamar grip dynamometer
VAS | 1 year
  Pain using the VAS (0-10)
DASH | 1 year
  Disabilities of the arm, shoulder and hand (0-100, lower score means better outcome)
PRWE | 1 year
  Patient rated wrist evaluation (0-100, lower score, means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lieselot Brepoels, MD, Study Director — RZ Tienen
Locations (1):
- Department of orthopaedics RZ Tienen, Tienen, Belgium

IPD SHARING:
Plan to Share IPD: No
clinical and economical data